CLINICAL TRIAL: NCT06331598
Title: A Phase II, Open Label, Randomized, Non-Comparative Cohorts Study of Adjuvant Atezolizumab or Atezolizumab Plus Tiragolumab in Solid Tumors with Resectable Disease with Intermediate-High Risk of Recurrence and High Tumor Mutational Burden (TMB-H) or Microsatellite Instability (MSI-H)
Brief Title: A Study of Adjuvant Atezolizumab or Atezolizumab Plus Tiragolumab in Solid Tumors with Resectable Disease with Intermediate-High Risk of Recurrence and High Tumor Mutational Burden (TMB-H) or Microsatellite Instability (MSI-H)
Acronym: IMperator
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Global desprioritization decision by the sponsor.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML43332; 2022-003708-33 (EudraCT Number)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atezolizumab (Experimental): Participants will be treated with atezolizumab every 4 weeks (Q4W) for 12 cycles (cycle = 28 days). After study treatment discontinuation participants will be followed until disease progression and afterwards, survival follow-up and new anti-cancer therapy will be collected until death (unless the participant withdraws consent, is lost to follow-up or the Sponsor terminates the study).
  Interventions: Drug: Atezolizumab
- Atezolizumab + Tiragolumab (Experimental): Participants will be treated with atezolizumab and tiragolumab Q4W for 12 cycles (cycle = 28 days). After study treatment discontinuation participants will be followed until disease progression and afterwards, information on survival follow-up and new anti-cancer therapy will be collected until death (unless the participant withdraws consent, is lost to follow-up or the Sponsor terminates the study).
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — A dose of 1680 mg atezolizumab will be administered intravenously on Day 1 of each 28-day cycle for a total of 12 cycles.
  Other Names: Tecentriq
Drug: Tiragolumab — A dose of 840 mg tiragolumab will be administered intravenously on Day 1 of each 28-day cycle for a total of 12 cycles.
  Other Names: MTIG7192A
  Arms: Atezolizumab + Tiragolumab

SUMMARY:
This study is being conducted to evaluate efficacy parameters (disease free survival [DFS] and overall survival [OS]) of atezolizumab and atezolizumab in combination with tiragolumab in TMB-H or MSI-H as adjuvant treatment after standard radical intended treatment in participants with intermediate-high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Any of the following solid tumors considered to be resectable with a curative intent: non-small cell lung cancer, skin melanoma, skin squamous cell carcinoma, urothelial carcinoma, colorectal cancer, gastric cancer, endometrial cancer, cervix cancer, head and neck cancer and any other tumor type with known high TMB (≥ 13 mut/MB) or MSI-H
* Participants must undergo standard treatment according to the stage of their disease and investigator´s choice
* All participants must be disease free after standard therapy to be included in this study
* Having TMB ≥ 13 mut/MB or MSI-H in tumor tissue biopsy obtained prior to starting standard treatment or from surgical specimens and analyzed using F1 CDx
* Participants must be at intermediate/high risk of recurrence
* Adequate hematologic and organ function
* Female participants of childbearing potential and male participants with female partners of childbearing potential must be willing to avoid pregnancy
* Women who are not postmenopausal or surgically sterile must have a negative serum pregnancy test result within 8 days prior to initiation of study drug.

Exclusion Criteria:

* Previous malignancies within 3 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Prior cancer immunotherapy
* Women who are pregnant, lactating, or intending to become pregnant during the study
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Significant cardiovascular disease
* Treatment with systemic immunosuppressive medications within 2 weeks prior to inclusion
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives of the drug, whichever is longer, prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2028-10-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) Rate at 24 Months | Month 24

SECONDARY OUTCOMES:
DFS Rate at 36, 48 and 60 Months | Months 36, 48, 60
OS (Overall Survival) | From randomization to death from any cause (up to approximately 60 months)
Percentage of Participants With Adverse Events | Up to approximately 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Spain (3):
  - Hospital Universitari Vall dHebron; Oncology, Barcelona, BARCELONA
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid, Madrid
  - Hospital Universitario Virgen; Servicio de Oncologia, Seville, SEVILLA

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing